CLINICAL TRIAL: NCT03277131
Title: A Prospective, Open, Non-Comparative Multicentre Study to Evaluate a Fibrous Silver Dressing (DURAFIBER™ Ag) in the Treatment of Moderate to Highly Exuding Venous Leg Ulcers
Brief Title: DURAFIBER Ag Post-Market Clinical Follow-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT1701DUR
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2020-06

CONDITIONS: Wounds and Injuries; Venous Leg Ulcer; Infection
MeSH Terms: conditions — Wounds and Injuries; Varicose Ulcer; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Antimicrobial Dressing
  Interventions: Device: DURAFIBER Ag

INTERVENTIONS:
Device: DURAFIBER Ag — DURAFIBER Ag is a commercially available absorbent, non-woven, silver-containing antimicrobial dressing

SUMMARY:
The aim of the study is to evaluate the performance of DURAFIBER Ag and to assess how many bacteria are present in infected wounds over an 8 week period.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the performance of DURAFIBER Ag and to assess how many bacteria are present in infected wounds over an 8 week period.

DURAFIBER Ag is a commercially available absorbent, non-woven, silver-containing antimicrobial dressing for use on a variety of exuding wounds and is widely used in routine clinical practice within the UK.

The primary outcome will be the quantitative reduction in bacterial load, based on a wound biopsy, from baseline to week 8. Secondary objectives will include the quantitative reduction in bacterial load, based on biopsy, from initial assessment to week 4, and the semi-quantitative reduction in bacterial load, based on swab analysis, from baseline to weeks 4 and 8. Additionally dressing performance measures will be assessed as well as all adverse events and device deficiencies.

In total 20 evaluable participants with an infected venous leg ulcer will be recruited into the trial. All participants will have their wound dressed using DURAFIBER Ag and will be followed-up for 8 weeks.

ELIGIBILITY:
Inclusion Criteria: Inclusion Criteria to be confirmed at the initial assessment

* The subject or must provide written informed consent.
* Subjects must be at least eighteen (18) years of age.
* Willing and able to make all required study visits.
* Able to follow instructions.
* Subjects must have a VLU, an ankle brachial pressure index (ABPI) taken within the last 28 days of 0.8-1.3, and must be treated with compression therapy.
* The subject must have a wound with an area ≥ 2cm².
* The subject's wound must have moderate or high exudate levels.
* The subject's reference wound must, in the opinion of the Healthcare Professional, show signs of infection warranting treatment with DURAFIBER Ag.
* In the clinician's opinion the subject's wound has an initial bacterial count of > 104 cfu/g (which will be confirmed following the initial wound biopsy).

Inclusion criteria to be confirmed when the biopsy result is recorded:

-The subject's wound has a confirmed initial bacterial count of > 104 cfu/g

Exclusion Criteria:

* Contraindications or hypersensitivity to the use of the DURAFIBER Ag, ancillary products or their components (e.g. known sensitivity to silver).
* Participation in the treatment period of another clinical trial within thirty (30) days of the date of consent.
* Subjects with skin features (e.g. tattoos, skin colour, pre-existing scarring) which, in the opinion of the Investigator, will interfere with the study assessments.
* Subjects receiving topical antimicrobials or oil-based products (such as petrolatum) at the reference wound surface.
* Subjects being treated with immunosuppressive drugs or corticosteroids.
* Subjects who have participated previously in this clinical trial and who have healed or been withdrawn.
* Subjects with a known history of poor compliance with medical treatment.
* Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Change in the mean log10 bacterial count in tissue biopsies from baseline to week 8 | 8 weeks

SECONDARY OUTCOMES:
Change in the mean log10 bacterial count from tissue biopsies from baseline to week 4. | 4 weeks
The semi-quantitative presence of bacteria, bacteria type and species from the weekly swabs | 8 weeks
Change in the number of subjects showing clinical signs of infection from baseline to weeks 4 and 8. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Helen Fearnley, Principal Investigator — Bradford Teaching Hospitals NHS Foundation Trust; Elizabeth Huddleston, PhD, Study Chair — Smith & Nephew - Global Strategy
Locations (7):
- United Kingdom (7):
  - Hull & East Riding Hospitals NHS Trust, Hull, East Yorkshire
  - Lancashire Care NHS Foundation Trust, Preston, Lancashire
  - Barnsley Hospital NHS Foundation Trust, Barnsley, South Yorkshire
  - Cardiff & Vale University Healthcare Board, Cardiff, Wales
  - Northumbria Healthcare NHS Foundation Trust, Ashington
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No